CLINICAL TRIAL: NCT04815031
Title: General Investigation of COMIRNATY Intramuscular Injection (Follow-up Study for Subjects [Healthcare Professionals] Who Are Vaccinated at an Early Post-Approval Stage)
Brief Title: Drug Use Investigation of COMIRNATY Intramuscular Injection
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591006
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
Keywords: COVID-19; Post-Marketing study, COMIRNATY,Vaccine
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COMIRNATY: COVID-19 mRNA vaccine (nucleoside-modified)
  Interventions: Biological: BNT162b2

INTERVENTIONS:
Biological: BNT162b2 — Comirnaty is administered intramuscularly after dilution as a course of 2 doses (0.3 mL each). It is recommended to administer the second dose 3 weeks after the first dose. Individuals 16 years of age and older.
  Other Names: COMIRNATY

SUMMARY:
Post-marketing study, Chotor study of COMIRNATY vaccenees followed for 11months. Serious adverse events and COVID-19 observed during the follow-up period will be collected, and the long-term safety of this product will be assessed.

DETAILED DESCRIPTION:
The healthcare professionals who are vaccinated with this product early after the marketing approval of this product (participants in the Investigation of Health Status of Recipients Vaccinated First conducted by the Science Research Group of the Ministry of Health, Labour and Welfare) will be followed for 11 months from the day following 28 days after the final vaccination of the initial immunization with this product (end date of observation period in Investigation of Health Status of Recipients Vaccinated First) to 12 months after the final vaccination of the initial immunization with this product, information on serious adverse events and COVID-19 observed during the follow-up period will be collected.

If booster vaccination isn't conducted, the long-term safety after the initial immunization of this product during the follow-up period will be assessed.

If booster vaccination is conducted, the long-term safety after the initial immunization of this product up to the day before booster vaccination will be confirmed, and information on serious adverse events and COVID-19 will be continuously obtained after booster vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have participated in the Investigation of Health Status of Recipients Vaccinated First and have provided written consent to continue participation in this study.

Exclusion Criteria:

* No exclusion criteria.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects who have been vaccinated with this product and have consented to participate in this study during participation in the Investigation of Health Status of Recipients Vaccinated First at contract sites.
Sampling Method: Probability Sample
Enrollment: 14570 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PfizerLocal Country Office, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591006

RESULTS

PARTICIPANT FLOW:
Groups:
- COMIRNATY Intramuscular Injection: The healthcare professionals who were vaccinated with this product early after the marketing approval of this product (participants in the Investigation of Health Status of Recipients Vaccinated First conducted by the Science Research Group of the Ministry of Health, Labour and Welfare) as indicated in the approved local product document were observed for a period of 11 months from the day following 28 days after the final vaccination of the initial immunization with this product to 12 months after the final vaccination of the initial immunization with this product.
  If booster vaccination was not conducted, the long-term safety after the initial immunization of this product during the follow-up period was assessed.
  If booster vaccination was conducted, the long-term safety after the initial immunization of this product up to the day before booster vaccination was confirmed, and information on serious adverse events and COVID-19 were continuously obtained after booster vaccination.
  This study only collected serious adverse events.
Period: Overall Study
Arm/Group | COMIRNATY Intramuscular Injection
Started | 14570
Received a Booster Vaccination in Completed Paticipants. | 13695 (Booster vaccination was not a condition of withdrawal. The number above shows the participant number who received a booster vaccination in the completed participants.)
Completed | 14537
Not Completed | 33
Not completed — No adverse event information (missing information) | 33

BASELINE CHARACTERISTICS:
Population: A total of 14570 participants were enrolled in this study. Of the 14570 participants from whom CRFs were collected, 33 participants were excluded from the safety analysis set due to no adverse event information (missing information).
Arm/Group | COMIRNATY Intramuscular Injection
Number analyzed (Participants) | 14537
Age, Customized [Number; unit: Participants]
  <15 years | 0
  ≥15 and <65 years | 14113
  ≥65 years | 424
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9744
  Male | 4793
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Serious Adverse Events
Description: A serious adverse event was any untoward medical occurrence resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; or congenital anomaly.
Time Frame: From the day following 28 days after the final vaccination of COMIRNATY, If those who did not conducted the booster vaccination was 11 months, If booster vaccination was conducted, up to the day before booster vaccination.
Population: The safety analysis set comprised of participants who satisfied the inclusion criteria and were vaccinated with COMIRNATY at least once. Participants with no adverse event information (missing information) were excluded.
Measure: Number; unit: Percentage of Participants
Groups:
- COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, up to the Day Before Booster: The healthcare professionals who were vaccinated with this product early after the marketing approval of this product (participants in the Investigation of Health Status of Recipients Vaccinated First conducted by the Science Research Group of the Ministry of Health, Labour and Welfare) as indicated in the approved local product document were observed for a period of 11 months from the day following 28 days after the final vaccination of the initial immunization with this product to 12 months after the final vaccination of the initial immunization with this product.
  If booster vaccination was not conducted, the long-term safety after the initial immunization of this product during the follow-up period was assessed.
  If booster vaccination was conducted, the long-term safety after the initial immunization of this product up to the day before booster vaccination was confirmed, and information on serious adverse events and COVID-19 were continuously obtained after booster vaccination.
  This study only collected serious adverse events.
Arm/Group | COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, up to the Day Before Booster
Number analyzed (Participants) | 14537
Percentage of Participants | 0.83

2. Primary Outcome: Proportion of Participants With Severe COVID-19
Description: By using the information on COVID-19 entered in the CRF submitted by the physician, participants who were considered to be in a severe condition were identified and the number and proportion of the participants were tabulated with reference to the severity classification in the Guidance for Treatment of Novel Coronavirus Infection (COVID-19).
  Participants with severe COVID-19 were defined as any of the following actions taken during the period from disease onset to the outcome date: admission to an ICU; use of mechanical ventilation; or use of ECMO.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, up to the Day Before Booster
Number analyzed (Participants) | 14537
Percentage of Participants | 0

3. Primary Outcome: Proportion of Participants With Serious Adverse Reactions
Description: A serious adverse reaction was any untoward medical occurrence attributed to COMIRNATY resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; or congenital anomaly. Relatedness to COMIRNATY was assessed by the physician.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, up to the Day Before Booster
Number analyzed (Participants) | 14537
Percentage of Participants | 0.03

4. Primary Outcome: Number of Participants With Serious Adverse Events After Booster Vaccination
Description: as for outcome 1
Time Frame: From the day of booster vaccination up to 11 months from the day following 28 days after the final vaccination of COMIRNATY. (out of scope of the safety evaluation)
Population: Participants who received booster vaccination regardless of COMIRNATY or other COVID-19 vaccines
Measure: Number; unit: Participants
Groups:
- COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, After the Booster: The healthcare professionals who were vaccinated with this product early after the marketing approval of this product (participants in the Investigation of Health Status of Recipients Vaccinated First conducted by the Science Research Group of the Ministry of Health, Labour and Welfare) as indicated in the approved local product document were observed for a period of 11 months from the day following 28 days after the final vaccination of the initial immunization with this product to 12 months after the final vaccination of the initial immunization with this product.
  If booster vaccination was not conducted, the long-term safety after the initial immunization of this product during the follow-up period was assessed.
  If booster vaccination was conducted, the long-term safety after the initial immunization of this product up to the day before booster vaccination was confirmed, and information on serious adverse events and COVID-19 were continuously obtained after booster vaccination.
  This study only collected serious adverse events.
Arm/Group | COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, After the Booster
Number analyzed (Participants) | 13695
Participants | 48

5. Primary Outcome: Number of Participants With Severe COVID-19 After Booster Vaccination
Description: as for outcome 2
Time Frame: as for outcome 4
Population: Participants who received booster vaccination regardless of COMIRNATY or other COVID-19 vaccines
Measure: Number; unit: Participants
Arm/Group | COMIRNATY (Tozinameran) ; If the Booster Vaccination Was Conducted, After the Booster
Number analyzed (Participants) | 13695
Participants | 0

6. Primary Outcome: Number of Participants With Serious Adverse Reactions After Booster Vaccination
Description: A serious adverse reaction was any untoward medical occurrence attributed to the vaccines received as a booster vaccination resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; or congenital anomaly. Relatedness to COMIRNATY was assessed by the physician.
Time Frame: as for outcome 4
Population: Participants who received booster vaccination regardless of COMIRNATY or other COVID-19 vaccines
Measure: Number; unit: Participants
Groups:
- COMIRNATY(Tozinameran);If the Booster Vaccination Was Conducted, After the Booster: The healthcare professionals who were vaccinated with this product early after the marketing approval of this product (participants in the Investigation of Health Status of Recipients Vaccinated First conducted by the Science Research Group of the Ministry of Health, Labour and Welfare) as indicated in the approved local product document were observed for a period of 11 months from the day following 28 days after the final vaccination of the initial immunization with this product to 12 months after the final vaccination of the initial immunization with this product.
  If booster vaccination was not conducted, the long-term safety after the initial immunization of this product during the follow-up period was assessed.
  If booster vaccination was conducted, the long-term safety after the initial immunization of this product up to the day before booster vaccination was confirmed, and information on serious adverse events and COVID-19 were continuously obtained after booster vaccination.
  This study only collected serious adverse events.
Arm/Group | COMIRNATY(Tozinameran);If the Booster Vaccination Was Conducted, After the Booster
Number analyzed (Participants) | 13695
Participants | 2

ADVERSE EVENTS:
Time Frame: From the day following 28 days after the final vaccination of COMIRNATY, If those who did not conducted the booster vaccination, the observation period was11 months, If booster vaccination was conducted, the obseravtion period was two types below. (1) Up to the day before booster vaccination. (2) After the booster vaccination. [From the day of booster vaccination up to the last day of observation period] (out of scope of the safety evaluation)
Description: Only serious adverse events were collected in this study. Other (not Including serious) adverse events were not assessed.
Groups:
- COMIRNATY (Tozinameran) (1) If the Booster Vaccination Was Conducted, up to the Day Before Booster.: The healthcare professionals who were vaccinated with this product early after the marketing approval of this product (participants in the Investigation of Health Status of Recipients Vaccinated First conducted by the Science Research Group of the Ministry of Health, Labour and Welfare) as indicated in the approved local product document were observed for a period of 11 months from the day following 28 days after the final vaccination of the initial immunization with this product to 12 months after the final vaccination of the initial immunization with this product.
  If booster vaccination was not conducted, the long-term safety after the initial immunization of this product during the follow-up period was assessed.
  If booster vaccination was conducted, the long-term safety after the initial immunization of this product up to the day before booster vaccination was confirmed, and information on serious adverse events and COVID-19 were continuously obtained after booster vaccination.
  This study only collected serious adverse events.
- COMIRNATY (Tozinameran) (2) If the Booster Vaccination Was Conducted, After the Booster.: Same as the left.
Arm/Group | COMIRNATY (Tozinameran) (1) If the Booster Vaccination Was Conducted, up to the Day Before Booster. | COMIRNATY (Tozinameran) (2) If the Booster Vaccination Was Conducted, After the Booster.
All-Cause Mortality (participants affected / at risk) | 1/14537 | 0/13695
Serious Adverse Events (participants affected / at risk) | 120/14537 | 48/13695
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | COMIRNATY (Tozinameran) (1) If the Booster Vaccination Was Conducted, up to the Day Before Booster. (N=14537) | COMIRNATY (Tozinameran) (2) If the Booster Vaccination Was Conducted, After the Booster. (N=13695)
Anaemia neonatal (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Prinzmetal angina (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Cleft lip (Congenital, familial and genetic disorders) | 1 | 0
Congenital skin disorder (Congenital, familial and genetic disorders) | 1 | 0
Gnathoschisis (Congenital, familial and genetic disorders) | 1 | 0
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 2 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 3 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial prostatitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
COVID-19 (Infections and infestations) | 9 | 15
Cystitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 3 | 0
Peritonsillitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 0
Airway burns (Injury, poisoning and procedural complications) | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 2
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Haemangioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 5 | 5
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 2 | 1
Cervical incompetence (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Placenta praevia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature labour (Pregnancy, puerperium and perinatal conditions) | 3 | 1
Dissociative disorder (Psychiatric disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 0
Ovarian cyst (Reproductive system and breast disorders) | 3 | 1
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Catamenial pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Respiratory disorder neonatal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Osteochondrodysplasia (Congenital, familial and genetic disorders) | 0 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT04815031/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT04815031/SAP_001.pdf